CLINICAL TRIAL: NCT00965965
Title: Effects of Comprehensibility of Colorectal Cancer Screening Educational Materials on Patient Knowledge and Motivation: A Randomized Controlled Trial
Brief Title: Comprehensibility of Colorectal Cancer Screening Educational Materials: Effects on Patient Knowledge and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Academy of Family Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 200917361-1
Record Dates: First submitted 2009-08-20; First posted 2009-08-26 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Colorectal Neoplasms
Keywords: health behavior; randomized controlled trials; self-efficacy; patient education; comprehension; mass screening; prevention and control
MeSH Terms: conditions — Colorectal Neoplasms; Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental patient education document (Experimental)
  Interventions: Behavioral: New colorectal cancer screening patient education document
- Traditional patient education document (Active Comparator)
  Interventions: Behavioral: Traditional colorectal cancer screening education document

INTERVENTIONS:
Behavioral: New colorectal cancer screening patient education document — The newly developed educational document was created accounting for health behavioral models (such as the Expanded Health Behavior Model, Social Cognitive Theory, and the Transtheoretical Model) and related research studies indicating the factors that most strongly and positively influence patients' cognitions regarding colorectal cancer screening and are, in turn, predictive of actual colorectal cancer screening behavior.
  Arms: Experimental patient education document
Behavioral: Traditional colorectal cancer screening education document — The traditional educational document is a slightly edited version of materials freely available on the National Cancer Institute (NCI) web site, used in this study with the permission of the NCI.
  Arms: Traditional patient education document

SUMMARY:
The purpose of this study is to determine whether a newly developed patient education document concerning colorectal cancer screening will be better understood and have greater effects on patient knowledge of and motivation for screening than a standard educational document.

ELIGIBILITY:
Inclusion Criteria:

* Receive primary care at one of the participating outpatient offices
* Age 50-75
* Able to read and speak English
* Adequate vision, hearing, and hand function to read printed documents, communicate with research staff, answer questionnaires, and otherwise participate
* Not up to date for colorectal cancer screening (defined as fecal occult blood test within 1 year, flexible sigmoidoscopy within 5 years, or colonoscopy within 10 years)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Comprehension of randomly assigned educational document | Immediately after receiving randomly assigned study intervention (that same day)

SECONDARY OUTCOMES:
Colorectal cancer screening knowledge | Immediately after receiving randomly assigned study intervention (that same day)
Self-efficacy for undergoing colorectal cancer screening | Immediately after receiving randomly assigned study intervention (that same day)
Perceived barriers to undergoing colorectal cancer screening | Immediately after receiving randomly assigned study intervention (that same day)
Readiness to undergo colorectal cancer screening | Immediately after receiving randomly assigned study intervention (that same day)

CONTACTS AND LOCATIONS:
Overall Officials: Tonantzin Rodriguez, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States